CLINICAL TRIAL: NCT04500457
Title: A Preliminary Evaluation of an Exposure-Based Treatment for Perfectionism
Brief Title: Exposure-Based Treatment for Perfectionism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jesse Cougle, Associate Professor of Psychology, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC2019.27351
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Perfectionism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm consists of a 2-week computerized, exposure-based intervention. Treatment sessions are completed every 3 days at home (5 treatment sessions total).
  Interventions: Behavioral: Exposure-based Treatment for Perfectionism (ETP)
- Wait-List Control (No Intervention): Participants in this condition will not receive treatment.

INTERVENTIONS:
Behavioral: Exposure-based Treatment for Perfectionism (ETP) — Three tasks focused on exposures are completed. Each treatment session is approximately twenty minutes.
  Arms: Intervention

SUMMARY:
This study is examining the efficacy of a computerized, exposure-based, intervention for perfectionism.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the effects of a two-week computerized exposure-based treatment for perfectionism (ETP). Individuals with elevated perfectionism will be randomly assigned to ETP or a waitlist (WL) control condition. ETP will consist of three tasks in which they will repeatedly make mistakes, repeated for five sessions over a two-week period (one session every 3 days).

ELIGIBILITY:
Inclusion Criteria:

* Score of at least 29 on the Frost Multidimensional Perfectionism Scale- Concern over Mistakes subscale

Exclusion Criteria:

* Current moderate or severe substance use disorder, psychotic disorder, or bipolar disorder
* Current suicidal ideation (imminent risk)
* Currently participating in psychotherapy
* Any changes to psychotropic medications in the past four weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Department of Psychology, Tallahassee, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Wait-List Control
Started | 39 | 37
Completed | 36 | 35
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Wait-List Control | Total
Number analyzed (Participants) | 39 | 37 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.10 (6.09) | 18.89 (1.31) | 19.91 (4.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 72
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 4 | 0 | 4
  White | 27 | 26 | 53
  Hispanic | 4 | 10 | 14
  Asian or Pacific Islander | 3 | 1 | 4
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 39 | 37 | 76

OUTCOME MEASURES:

1. Primary Outcome: Frost Multidimensional Perfectionism Scale (FMPS)- Concern Over Mistakes Subscale
Description: Self-report questionnaire examining levels of perfectionism. The concern over mistakes sub-scale of the Frost Multidimensional Perfectionism Scale includes 9 items with scores on the sub-scale ranging from 9 to 45 (higher scores signify higher levels of concern over mistakes). The concern over mistakes sub-scale includes the following items from the Frost Multidimensional Perfectionism Scale: 9, 10, 13, 14, 18, 21, 23, 25, 24. Item scores are summed for a total sub-scale score.
Time Frame: Levels of perfectionism from baseline to post treatment (2 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Wait-List Control
Number analyzed (Participants) | 36 | 35
units on a scale
  Baseline | 36.54 (4.10) | 35.76 (4.06)
  Post-test | 30.97 (6.39) | 35.71 (4.16)

2. Secondary Outcome: Center for Epidemiological Studies Depression Scale (CES-D)
Description: Self-report measure used to assess depressive symptoms. Total scores range from 0 to 60 with higher scores indicating a higher level of depressive symptoms.
Time Frame: Depression symptoms from baseline to post treatment (2 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Wait-List Control
Number analyzed (Participants) | 36 | 35
units on a scale
  Baseline | 19.26 (8.33) | 22.97 (12.75)
  Post-test | 14.69 (8.12) | 23.77 (11.47)

3. Secondary Outcome: State-Trait Inventory for Cognitive and Somatic Anxiety-Trait Version (STICSA-T)
Description: Self-report measure used to assess overall anxiety symptoms. Scores range from 21 to 84 with higher scores indicating higher levels of overall anxiety.
Time Frame: Anxiety symptoms from baseline to post treatment (2 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Wait-List Control
Number analyzed (Participants) | 36 | 35
units on a scale
  Baseline | 41.33 (9.75) | 43.95 (12.90)
  Post-test | 39.19 (11.07) | 43.95 (11.10)

4. Secondary Outcome: Social Phobia Inventory (SPIN)
Description: Self-report scale that measures Social anxiety symptoms. Scores range from 0 to 68 with higher scores indicating higher levels of social anxiety symptoms.
Time Frame: Social anxiety symptoms from baseline to post treatment (2 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Wait-List Control
Number analyzed (Participants) | 36 | 35
units on a scale
  Baseline | 29.15 (13.08) | 30.08 (17.12)
  Post-test | 26.58 (12.79) | 32.31 (16.36)

5. Secondary Outcome: Eating Attitudes Test (EAT-26)
Description: Self-report scale that measures eating disorder symptoms. Scores range from 0 to 78 with higher scores indicating higher levels of eating disorder symptoms.
Time Frame: Eating disorder symptoms from baseline to post treatment (2 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Wait-List Control
Number analyzed (Participants) | 36 | 35
units on a scale
  Baseline | 13.82 (9.09) | 12.03 (9.63)
  Post-test | 12.05 (9.46) | 14.34 (11.18)

6. Secondary Outcome: Obsessive-Compulsive Inventory- Revised (OCI-R)
Description: Self-report scale that measures obsessive-compulsiveness. Scores range from 0 to 72 with higher scores indicating higher levels of obsessive-compulsiveness.
Time Frame: Obsessive-compulsiveness from baseline to post treatment (2 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Wait-List Control
Number analyzed (Participants) | 36 | 35
units on a scale
  Baseline | 22.89 (13.18) | 26.68 (13.67)
  Post-test | 21.34 (13.95) | 25.54 (13.24)

ADVERSE EVENTS:
Time Frame: Baseline up to 2 weeks
Arm/Group | Intervention | Wait-List Control
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/37
Other Adverse Events (participants affected / at risk) | 0/39 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT04500457/Prot_SAP_000.pdf